CLINICAL TRIAL: NCT06149858
Title: Ventral Mesh Hernioplasty : Laparoscopic Versus Open Sublay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed hussein abozeid ahmed, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ventral hernia repair
Record Dates: First submitted 2023-11-10; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral | interventions — Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sublay (Experimental): patients with ventral hernia operated as sublay mesh repair positioning of mesh under sheath
  Interventions: Procedure: hernioplasty
- laparoscopic (Experimental): patients with ventral hernia operated as laparoscopic repair positioning TAPP mesh
  Interventions: Procedure: hernioplasty

INTERVENTIONS:
Procedure: hernioplasty — ventral hernia repair with mesh

SUMMARY:
To compare between laparoscopic ventral hernia repair and open sublay technique (recurrence ,operative time ,bleeding ,rate of complication and injury , seroma, post operative pain)

DETAILED DESCRIPTION:
A hernia usually happens in abdomen or groin, when one of your organs pushes through the muscle or tissue that contains it. Most hernias eventually will need surgical repair.

sublay mesh repair has the lowest recurrence and surgical site infection in open anterior abdominal hernia repair it is a perfect choice for the repair of ventral abdominal hernia the principles included two main steps: (1) mesh placement deep into the recti muscles and (2) mesh extension beyond the hernia defect.

Laparoscopic ventral hernia repair (LVHR) has established itself as a well-accepted option in the treatment of hernias. Clear benefits have been established regarding the superiority of LVHR in terms of fewer wound infections compared with open repairs. Meticulous technique and appropriate patient selection are critical to obtain the reported results.

• In the laparoscopic technique, a prosthetic mesh is inserted through a trocar into the abdominal cavity and fixed against the abdominal wall. After reducing the hernia contents, the hernia sac is left unresected, and most surgeons do not place additional sutures for closing the hernia orifice. A specific risk of laparoscopic hernia repair lies in freeing adhesions between intestine and abdominal wall, which may result in (sometimes unrecognised) bowel perforation . The mesh should overlap the hernia orifice by at least 5 cm and is anchored to the abdominal wall with tacks, transfascial sutures, or a combination of the two methods. In laparoscopic abdominal hernia repair, mesh placement methods are generally classified into intraperitoneal onlay mesh (IPOM), transabdominal abdominal preperitoneal (TAPP)

ELIGIBILITY:
Inclusion Criteria:

* All cases of midline ventral hernia fit for surgery

Exclusion Criteria:

1. Surgically unfit cases
2. Complicated hernia (obstructed ,irreducible, strangulated)
3. incisional ,massive ,recurrent hernias

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | baseline
  compare between laparoscopic ventral hernia repair and open sublay technique in how long the hernia take to occur again

CONTACTS AND LOCATIONS:
Overall Officials: hisham ryad, Study Director

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Issa M, Noureldin K, Elgadi A, Abdelaziz A, Badawi M, Makram M. Evaluation of the Sublay Mesh Repair Outcomes in Different Types of Ventral Hernia. Cureus. 2021 Dec 21;13(12):e20590. doi: 10.7759/cureus.20590. eCollection 2021 Dec. PMID 35103166